CLINICAL TRIAL: NCT00220259
Title: Cystic Fibrosis Withdrawal of Inhaled Steroids Evaluation Study (CF WISE Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Cystic Fibrosis Trust (Other); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01PRT/31; Cystic Fibrosis Trust; PJ498
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2005-11-08 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis, inhaled corticosteroids
MeSH Terms: conditions — Cystic Fibrosis | interventions — Fluticasone

INTERVENTIONS:
Drug: Fluticasone or placebo

SUMMARY:
The overall aim of this study is to find out whether taking regular inhaled steroids (eg Pulmicort, Flixotide, Becotide, Becloforte) is good for the lungs of children and adults with cystic fibrosis (CF).

Some patients are put on inhaled steroids because they are wheezy despite taking regular bronchodilators (inhaled medicines that help open up the airways eg Ventolin, Bricanyl). Occasionally young children are put on them when they wheeze with colds, and have simply remained on them ever since. However many CF patients have been put onto inhaled steroids because their doctors thought it might reduce the inflammation in the lungs and help improve lung function. This inflammation (which is swelling of the lining of the airways) is known to be important in CF and results from recurrent chest infections.

Although it is believed, in theory, that inhaled steroids should be useful for most CF patients, we are not sure how well they work in CF and it has not yet been possible to prove this with standard studies. This would normally involve starting inhaled steroids in patients who have not been taking them. We have therefore taken a different approach, namely to withdraw them from some patients who have been on them for a long time, to see if there is any effect of stopping them.

It is important that we answer this question, as we do not want CF patients taking medicines that may be unnecessary. CF patients already have to take many oral and inhaled medicines and if we can cut down this burden, it would be helpful for everyone. Of course, we may find that patients do need these medicines but at least we will then be certain that it is for a good reason.

The main hypothesis is that withdrawing inhaled steroids is not associated with an earlier onset of acute chest exacerbations.

DETAILED DESCRIPTION:
Background: Long term, and often high dose, inhaled corticosteroids (ICS) are being increasingly prescribed to patients with CF to combat lung inflammation. Despite five published studies, a Cochrane systematic review has concluded that there is not enough evidence of either benefit or harm. The number of CF patients already taking ICS in the UK means recruitment into conventional studies has proved difficult.

Aims: to test the feasibility and safety of withdrawal of ICS in CF by performing a study of randomised placebo-controlled withdrawal of ICS in children and adults already taking them. The results will be used to determine the feasibility of a future prospective study to prove whether starting ICS in CF patients not already on them, and those successfully withdrawn, leads to benefit (in lung function and chest exacerbations) and/or harm, compared to placebo.

Methods: We will study 240 children and adults in 12 centres. We have matching placebo and Flixotide metered dose inhalers to be used through a Volumatic, so any subjects currently on Pulmicort or Becotide will switch to Flixotide 2 months during the run-in phase, and all subjects will use their ICS through a spacer device. Patients will be randomised to continue on ICS or take placebo for 6 months, in a double-blind fashion. Primary outcome is time to 1st exacerbation; secondary ones are decline in lung function, new courses of antibiotics and rescue bronchodilator usage.

ELIGIBILITY:
Inclusion Criteria:

.Diagnosis of CF (positive sweat test or DNA analysis). .Age over 6.0 years (no upper limit). .FEV1 > 40% predicted for gender, height and age. .Already taking ICS for at least 3 months. .Patients who are able to perform spirometry and can correctly use their prescribed inhaler.

.Patients whose parents or legal guardians are willing to give written informed consent for their child to participate in the study. The investigators will also obtain consent from the child whenever possible.

.Patients who are likely to cooperate with taking the study medication and attend the clinic at appointed times.

Exclusion Criteria:

* Taking oral corticosteroids, usually for allergic bronchopulmonary aspergillosis (ABPA), currently or within the previous month.
* Cases in which the clinician feels unhappy about stopping ICS due to severe lung disease or concomitant "asthma" (see below).
* Course of intravenous antibiotics (IVABs) within last month.
* Taking part in another drug trial within last 2 months. .Use of high doses of inhaled corticosteroids (greater than or equal to 2000mcg/d fluticasone for 17 years or over and greater than or equal to 1000mcg/d fluticasone if less than 17 years.
* Patients with any medical or psychological condition, which in the opinion of the investigators precludes their entry into the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 2001-05; Study Completion 2005-02

PRIMARY OUTCOMES:
Time to first respiratory exacerbation

SECONDARY OUTCOMES:
Decline in lung function
New courses of antibiotics
Bronchodilator usage

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Balfour Lynn, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, London, United Kingdom